CLINICAL TRIAL: NCT02878031
Title: Community Case Management of Chest Indrawing Pneumonia With Oral Amoxicillin in Children Aged 2-59 Months Old by Community Oriented Resources Persons (CORPs) in Niger State, Nigeria
Brief Title: Community Case Management of Chest Indrawing Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Malaria Consortium (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HQGMP1611887
Record Dates: First submitted 2016-08-17; First posted 2016-08-25 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Pneumonia
Keywords: Integrated Community Case Management; Community Health Worker; Nigeria
MeSH Terms: conditions — Pneumonia | interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral amoxicillin for CI pneumonia (Experimental): Community management of chest indrawing pneumonia using oral amoxicillin by CHWs
  Interventions: Drug: Oral amoxicillin for CI pneumonia

INTERVENTIONS:
Drug: Oral amoxicillin for CI pneumonia — CHW management of chest indrawing (CI) pneumonia in children 2-59 months old using oral amoxicillin, given in the following age specific dosage:
  2 months ≤ children age <12 months (4 - <10kg): one (1) tablet 250mg dispersible amoxicillin twice daily (morning and evening) for 5 days.
  12 months≥ children age <3 years (10 kg - <14 kg): two (2) tablets 250mg dispersible amoxycillin taken twice daily (morning and evening) for 5 days.
  ≥ 3 years of age children <5 years (14kg - 19kg): three (3) tablets 250mg dispersible amoxycillin taken twice daily (morning and evening) for 5 days.
  Other Names: Intervention arm

SUMMARY:
This one-arm safety intervention study is aimed at increasing access to treatment of pneumonia by training CHWs, locally referred to as Community Oriented Resource Persons (CORPs), to manage chest indrawing pneumonia using oral amoxicillin, conducting follow-ups and recording their findings in case report forms. CORPs will also be involved in improving care seeking for pneumonia in children by training them to conduct health education sessions for men and women in their respective communities.

The primary objective is to assess if CORPs can safely and appropriately manage chest indrawing pneumonia in 2-59 month old children, and refer children with danger signs. The primary outcomes will be the proportion of children under five with chest indrawing pneumonia who were managed appropriately by CORPs and the clinical treatment failure of chest indrawing pneumonia. Secondary outcomes will include proportion of children with chest indrawing followed up by CORPs on day 3 and caregiver adherence to treatment for CI, and clinical relapse of pneumonia between day 7 to 14 among children whose signs of pneumonia disappeared by day 6. Approximately 308 children 2-59 months of age with chest indrawing pneumonia would be needed for this safety intervention study.

DETAILED DESCRIPTION:
OBJECTIVES AND RATIONALE This one-arm safety intervention study aims to establish whether CHWs in Nigeria can safely manage chest indrawing pneumonia in 2-59 month old children. The primary outcomes will be the proportion of children under five with chest indrawing pneumonia who were managed appropriately by Community Oriented Resources Persons (CORPs) and the clinical treatment failure by day 6. Secondary outcomes will include proportion of children with chest indrawing followed up by CORPs on day 3, clinical relapse of pneumonia between day 7 to 14 and acceptability and satisfaction with outpatient management of chest indrawing pneumonia. A total of 308 children 2-59 months of age with chest indrawing pneumonia will be needed for this safety intervention study.

EXPERIMENTAL DESIGN AND METHODOLOGY Introduction Malaria Consortium (MC) intends to implement the WHO study, funded under the Rapid Access Expansion 2015 programme (RAcE 2015), on community case management of chest indrawing pneumonia with oral amoxicillin in children aged 2-59 months old by CORPs and submits this proposal for Niger state, Nigeria.

Study area Proposed study population Niger State, located in Nigeria's North Central Zone, is geographically the largest of the country's states, covering 76,263 km2. The state has a projected population of almost 5 million. Children under five years make up 21% of the population, and pregnant women constitute 5%. The population is made up of Muslims, Christians with a small minority practising traditional beliefs. The majority of the population are spread across rural areas, with 30% of the population living in urban areas. Under WHO RAcE 2015 project MC is working with the Federal Ministry of Health (FMoH) to strengthen the iCCM programme in six (LGAs) in the three zones in Niger state: Paikoro; Rafi; Mariga; Rijau; Lapai; and Edati. The total population of the six LGAs is 1,245,939 of whom approximately 249,200 are children aged 2-59 months. Pneumonia remains the leading cause of under 5 child mortality in Nigeria which, together with India, contributes the highest absolute numbers of pneumonia deaths in the world, with 804,429 deaths in children under five years in 2013 (2). The expected incidence of clinical pneumonia in this area in Nigeria is 0.28/child/year with an estimated 12% progressing to severe disease.

Objectives and outcomes This one-arm safety intervention study aims to establish whether CHWs in Nigeria can safely and appropriately manage chest indrawing pneumonia in 2-59 month old children.

Primary outcomes will be the proportion of children under five classified with chest indrawing pneumonia who were managed appropriately by Community Oriented Resources Persons (CORPs) and the clinical treatment failure of chest indrawing pneumonia by day 6.

Secondary outcomes will include:

* Proportion of children classified with chest indrawing who were followed up by the CORPs on day 3
* Clinical relapse of pneumonia between day 7 to 14 among children whose signs of pneumonia disappeared by day 6
* CORPs' acceptability of and caregiver satisfaction with outpatient management of chest indrawing pneumonia

Sample size and sampling Using the sample size calculation for a prevalence survey with finite population correction; an assumption that the proportion of the main indicator is 50% (to give the most conservative sample size); and a confidence interval of 95%, a total of 196 children with chest indrawing will be needed to estimate overall proportion of children with chest indrawing pneumonia who experience treatment failure by day 6 with ±7% precision. Adjusting for a 10% non-response rate for caregivers, 10% erroneous enrolments, and a cluster effect of 1.3 in case more than one child is enrolled by one CORP, a total sample size of 308 children under five with chest indrawing will be required. After 12 months of data collection, an interim analysis of the event rates (primary outcome) and enrolment rates is planned to assess progress towards the sample size target. Should it be discovered that the event rate is far off from the assumption of 0.5, the final sample size may be modified.

With approximately 28,000 children 2-59 months old in the study area, assuming 7,840 fast breathing cases per year (0.28 episodes/child/year), and a 12% chest indrawing incidence the area would have approximately 940 chest indrawing cases per year. To enrol the 308 children with chest indrawing needed for the study during a 12 months study period we would need all the 203 CORPs in the LGA to see approximately 30% of the sick children in the community, which we believe is highly feasible given our experience with iCCM programmes uptake in other parts of Africa and the fact that we shall implement community mobilisation activities to support engagement with the study.

Case identification by CORPs will be mainly through passive case detection and through periodic community outreach activities. Based on epidemiological data, over a period of study data collection of 12 months maximum, each CORP is anticipated to enrol 1-2 children with chest indrawing. CORPs will assess all children presenting to their house and manage them according to study protocol. All sick infants younger than 2 months will be referred to the reference facility. All children 2-59 months of age with chest indrawing but no danger signs will be considered eligible for enrolment in the study and consent will be obtained from the primary caregiver. CORPs will screen the children for study enrolment, and takes consent from the guardian of the child to take part in the study. If the caregiver of the eligible child has consented, the CORP prescribes dispersible amoxicillin according to age-specific standards, schedules follow-up visits for day 0 (<12hrs), 3, 6 and 15 with caregiver of enrolled child, attaches a unique identifier (UI) to the sick child recording form of enrolled child and copies the UI number onto all copies of the consent form and gives a missed call to the RA to notify them of enrolled child.

The RA will visit the household of the child as soon as possible after the child has been enrolled and latest within 12 hours of enrolment by the CORP. Before going to the child's household, the RA will go to the CORP to verify the enrolment and get details of the child's location. The CORP will visit the child three days after enrolment (day 3) to ensure there is no deterioration in the child's condition and if necessary, refer the child to a health facility if symptoms have deteriorated. On day 6 and 15 after enrolment, RAs together with CORPs will visit all children enrolled and interview the caregivers using a mobile phone data collection form. Clinical relapse of pneumonia will be determined based on child's clinical condition assessed on day 15 (see table 4 for detailed definition of primary and secondary outcomes). If on any of the follow-up days, enrolled children cannot be found at home, the CORP/RA will follow up with the caregiver to find out where the child is, and make every effort to see the child, even if they are classified as lost to follow-up.

Data collection, supervision and outcome assessment

DAY 1:

The CORPs' performance will be established through a re-assessment of the child by a research assistant (RA) who will visit the household of the child as soon as possible after the child has been enrolled and latest within 12 hours of enrolment by the CORP. The RA will use a tablet based sick child assessment tool which walks the RA through questions about the child, including current health status and symptoms present at the time of care seeking at the CORPs, treatment given by CORP, and other treatments provided for the current illness episode. A handheld pulse oximeter will be used by the RAs to detect symptoms of hypoxemia. If a child is found to have danger signs or hypoxemia, or any other illness that was not treated by the CORP, the RA will facilitate referral to the nearest health facility and will be excluded from the study. For children with chest indrawings referred by the CORPs because of suspected presence of danger signs, the RA will trace the child in the referral facility (or at home in case of referral refusal) to conduct the re-assessment visit. Children found not to have chest indrawing will continue the course of antibiotic they were already prescribed.

DAY 3:

Families of enrolled children will be encouraged to return to the CORPs on 3 days after enrolment for reassessment by the CORP, as is standard under iCCM. During the this visit, the CORP will reassess the child, record findings (including temperature and presence/absence of chest indrawing and other treatments, if any, received by the child), inquire and record if the caretaker provided the amoxicillin tablets according to the recommended treatment schedule, and counsel the mother to administer the next doses. If a child is not brought back on the scheduled visit day, the CORP will visit the child at home on day 3 and 6. If the CORP determines that the condition of an enrolled child has deteriorated, s/he will refer the child to the reference facility or call the supervisor for further evaluation. Data on a standard set of variables will be collected during each visit. The study supervisors will verify that visits are being made and information is being collected by reviewing data uploads on the back-end server.

DAYS 6-15:

On day 6 and 15 after enrolment, RAs and CORPs will visit all children enrolled and interview the caregivers using the mobile phone data collection form. Questions will include current health status (using the IMCI algorithm), adherence to treatment (using pill count), care providers visited after visiting the CORP, alternative treatments given (other than what CORP provided), and hospitalisation. Clinical relapse of pneumonia will be determined based on child's clinical condition assessed on day 15. If enrolled children cannot be found at home during the day 6 and day 15 visits, the RA will follow up with a phone call to the caregiver to ensure that there is no loss-to follow-up.

Following the household visits on day 6 and 15, a selection of 25 CORPs and 25 child caregivers will be asked to participate in unstructured interviews to document CORPs' acceptability of and caregiver satisfaction with outpatient management of chest indrawing pneumonia.

The study coordinator will visit all of the treatment failures (secondary outcome) for reassessment of the child.

Monitoring and evaluation, including a summary of the data analysis plan A system for regular monitoring will be introduced to ensure that study activities are implemented as per plan, using approved operating procedures. CORP service statistics on patients seen and referrals made will be captured from both CORPs paper-based reports. This data will be compiled by a data manager, interpreted by the study coordinator and shared with program managers on a regular basis. The data manager will regularly review all data submissions for enrolled children, including checklists submitted by RAs on Day 0-1, 6 and 15, as well as follow-up forms submitted by CORPs on day 3. These submissions will be checked for completeness and accuracy before being anonymised by assigning each enrolled child a unique study number and using this number to store the case data in a project database. While all data collection forms will have inbuilt consistency and range checks, any additional discrepancies identified will be raised during supervision visits. An automatically generated report containing information on children enrolled, children followed up and children who died, had clinical treatment failure or who had a clinical relapse of pneumonia will be generated for review on a monthly basis and be made available to the PIs, co-investigators and the donor.

ELIGIBILITY:
Inclusion Criteria:

- Chest indrawing pneumonia

Exclusion Criteria:

* Convulsions
* Cough for 14 days or more
* Blood in stool
* Fever for last 7 days or more
* Diarrhoea for 14 days or more
* Not able to drink or feed anything
* Unusually sleepy or unconscious
* Vomits everything
* Swelling of both feet
* Red on MUAC strap (severe acute malnutrition)

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 191 (Actual)
Dates: Start 2016-10; Primary Completion 2018-05-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinical treatment failure | By day 3 to 6
  The proportion of children enrolled with any of the following signs by day 6:
  * Appearance of a danger sign (unable to drink or breastfeed, convulsions, vomiting after ingestion of food or drink, and abnormally sleepy or difficult to wake)
  * Hypoxemia (Oxygen saturation ≤90%)
  * Temperature ≥37.5°C and chest indrawing on day 3
  * Temperature ≥37.5°C or chest indrawing alone on day 6
  * Change of antibiotic
  * Death
Number of CHWs appropriately managing chest indrawing pneumonia | At day of enrolment
  Proportion of children with RA verified chest indrawing pneumonia with no referral sign (unable to drink or breastfeed, convulsions, vomiting after ingestion of food or drink, and abnormally sleepy or difficult to wake, malnutrition) who received the correct age-specific amoxicillin dose for 5 days Proportion of children with RA verified chest indrawing pneumonia with suspected referral sign (unable to drink or breastfeed, convulsions, vomiting after ingestion of food or drink, and abnormally sleepy or difficult to wake, malnutrition) who were given pre-referral amoxicillin treatment and were referred to a health facility.

SECONDARY OUTCOMES:
Number of children with chest indrawing pneumonia followed up by CHWs | By day 3
  The proportion of children enrolled with chest indrawing pneumonia who were seen and reassessed by a CHW 3 days after the initial visit
Number of children with clinical relapse of pneumonia | Between day 7 and 15
  The proportion of children enrolled who were clear of pneumonia symptoms (fast breathing and chest indrawing) on the day 6 visit with any of the following on day 15:
  * Appearance of any danger sign (as per above)
  * Chest indrawing
  * Fever ≥37.5°C
  * Fast breathing (as per WHO definition)
Number of caregivers who find outpatient management of chest indrawing pneumonia acceptable for their child | 15 days after enrolment
  The proportion of children enrolled whose caregivers administered a correct daily dose of antibiotics for the correct frequency and duration

CONTACTS AND LOCATIONS:
Overall Officials: Karin Kallander, MSc, PhD, Principal Investigator — Malaria Consortium; Ebenezer Baba, MD, MPH, Principal Investigator — Malaria Consortium
Locations (1):
- Piakoro & Lapai Local Government Areas, Minna, Niger State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
The DSMB will review all documents provided to the DSMB as well as all anonymised patient data
  * To review the conduct of the study, including protocol violations
  * To review data on participant recruitment, accrual, and retention, as well as assessments of data quality, completeness, and timeliness
  * Protect the confidentiality of the study data and the DSMB discussions
  * To make recommendations to continue, modify, or terminate the study depending upon these analyses
  * Operate according to the procedures described in this charter and all procedures of the DSMB.

REFERENCES:
- [Background] Countdown to 2015. Fulfilling the Health Agenda for Women and Children: The 2014 Report. World Health Organization and UNICEF, 2013.
- [Background] Liu L, Oza S, Hogan D, Perin J, Rudan I, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of child mortality in 2000-13, with projections to inform post-2015 priorities: an updated systematic analysis. Lancet. 2015 Jan 31;385(9966):430-40. doi: 10.1016/S0140-6736(14)61698-6. Epub 2014 Sep 30. PMID 25280870
- [Background] Kallander K, Hildenwall H, Waiswa P, Galiwango E, Peterson S, Pariyo G. Delayed care seeking for fatal pneumonia in children aged under five years in Uganda: a case-series study. Bull World Health Organ. 2008 May;86(5):332-8. doi: 10.2471/blt.07.049353. PMID 18545734
- [Background] Noordam AC, Carvajal-Velez L, Sharkey AB, Young M, Cals JW. Care seeking behaviour for children with suspected pneumonia in countries in sub-Saharan Africa with high pneumonia mortality. PLoS One. 2015 Feb 23;10(2):e0117919. doi: 10.1371/journal.pone.0117919. eCollection 2015. PMID 25706531
- [Background] Sazawal S, Black RE; Pneumonia Case Management Trials Group. Effect of pneumonia case management on mortality in neonates, infants, and preschool children: a meta-analysis of community-based trials. Lancet Infect Dis. 2003 Sep;3(9):547-56. doi: 10.1016/s1473-3099(03)00737-0. PMID 12954560
- [Background] Gupta GR. Tackling pneumonia and diarrhoea: the deadliest diseases for the world's poorest children. Lancet. 2012 Jun 9;379(9832):2123-4. doi: 10.1016/S0140-6736(12)60907-6. No abstract available. PMID 22682449
- [Background] Peterson S, Nsungwa-Sabiiti J, Were W, Nsabagasani X, Magumba G, Nambooze J, Mukasa G. Coping with paediatric referral--Ugandan parents' experience. Lancet. 2004 Jun 12;363(9425):1955-6. doi: 10.1016/S0140-6736(04)16411-8. PMID 15194257
- [Background] Kallander K, Tomson G, Nsungwa-Sabiiti J, Senyonjo Y, Pariyo G, Peterson S. Community referral in home management of malaria in western Uganda: a case series study. BMC Int Health Hum Rights. 2006 Mar 16;6:2. doi: 10.1186/1472-698X-6-2. PMID 16539744
- [Background] Walker CLF, Rudan I, Liu L, Nair H, Theodoratou E, Bhutta ZA, O'Brien KL, Campbell H, Black RE. Global burden of childhood pneumonia and diarrhoea. Lancet. 2013 Apr 20;381(9875):1405-1416. doi: 10.1016/S0140-6736(13)60222-6. Epub 2013 Apr 12. PMID 23582727
- [Result] Bari A, Sadruddin S, Khan A, Khan Iu, Khan A, Lehri IA, Macleod WB, Fox MP, Thea DM, Qazi SA. Community case management of severe pneumonia with oral amoxicillin in children aged 2-59 months in Haripur district, Pakistan: a cluster randomised trial. Lancet. 2011 Nov 19;378(9805):1796-803. doi: 10.1016/S0140-6736(11)61140-9. Epub 2011 Nov 10. PMID 22078721
- [Result] Soofi S, Ahmed S, Fox MP, MacLeod WB, Thea DM, Qazi SA, Bhutta ZA. Effectiveness of community case management of severe pneumonia with oral amoxicillin in children aged 2-59 months in Matiari district, rural Pakistan: a cluster-randomised controlled trial. Lancet. 2012 Feb 25;379(9817):729-37. doi: 10.1016/S0140-6736(11)61714-5. Epub 2012 Jan 27. PMID 22285055